CLINICAL TRIAL: NCT00653263
Title: Characterizing Methamphetamine Withdrawal in Recently Abstinent Methamphetamine Users: A Pilot Study
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 51178; Alcohol & Substance Dependence (Other: Other)
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Results first posted 2010-03-09 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2010-02

CONDITIONS: Methamphetamine Dependence; Methamphetamine Withdrawal
Keywords: methamphetamine; drug abuse; withdrawal
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Methamphetamine dependent: Methamphetamine dependent participants admitted to Recovery Centers of Arkansas

SUMMARY:
Methamphetamine use has escalated in recent years. Methamphetamine use has also spread throughout the country. Although much information has been gathered on the treatment of cocaine abuse, very little information has been obtained on the treatment of methamphetamine abuse. One of the first steps in developing appropriate treatment is to examine the effects of stopping a particular substance's use on individuals abusing that substance. To date this has not been well studied for people abusing methamphetamine. The purpose of this study is to better understand and develop accurate ways of measuring symptoms associated with stopping the use of methamphetamine in people that are abusing methamphetamine. If the withdrawal symptoms are able to be effectively measured, this will help to develop treatments targeted at alleviating these symptoms. These symptoms are often associated with relapse to use of that substance.

DETAILED DESCRIPTION:
The primary aim of this 4 week observational study is to examine and characterize the withdrawal symptoms experienced by methamphetamine abusers who are recently abstinent from methamphetamine. The period of drug or substance withdrawal is often cited as the time during which risk of relapse use of that substance is very high. Therefore it is highly important to characterize specifically the withdrawal syndrome associated with cessation of methamphetamine use. This study will demonstrate our ability to recruit and work with this methamphetamine dependent population. In addition it will allow for the collection of pilot data to assist in selecting appropriate assessment tools in a submission of an RO1 grant for well-controlled studies characterizing methamphetamine withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Subjects must have a history of methamphetamine use, with recent use verified by a urine toxicology screen positive for amphetamines

Exclusion Criteria:

* Current diagnosis of drug or alcohol physical dependence (other than methamphetamine or tobacco)
* Schizophrenia, or bipolar type I disorder
* Present or recent use of over-the-counter or prescription psychoactive drug or drug(s) that may affect mood ratings
* Current suicidality or psychosis
* Pregnancy: hormonal changes during pregnancy can affect mood which might produce a potential confound if pregnant women were enrolled

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll 20 methamphetamine dependent individuals ages 18-65 recruited from those admitted to the Recovery Centers of Arkansas in North Little Rock.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2006-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Mancino, M.D., Principal Investigator — University of Arkansas; Alison Oliveto, PhD, Study Chair — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 13 participants were recruited for enrollment in study entry.
Pre-assignment Details: A total of 5 participants did not meet study criteria and did not enter the study proper, leaving a total of 8 eligible subjects.
Period: Overall Study
Arm/Group | Methamphetamine Dependent
Started | 8 (1 dropped out of treatment and the other had untreated hypertension)
Completed | 6
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Methamphetamine Dependent
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.67 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Methamphetamine Selective Severity Assessment (MSSA)
Description: Methamphetamine Selective Severity Assessment (MSSA) is an 18 item questionnaire assessing withdrawal symptoms with each question measured on a scale from 0(best score)-7(worst score) for a range in scores from 0(best score)-126(worst score). Higher scores indicate more severe withdrawal symptoms.
Time Frame: Baseline through week 4
Measure: Mean (Standard Deviation); unit: "units on a scale"
Arm/Group | Methamphetamine Dependent
Number analyzed (Participants) | 6
"units on a scale" | 48.2 (26.8)
Statistical Analysis 1: Comparison: Methamphetamine Dependent; Means and ranges were computed for the continuous baseline characteristics.For data with 5 time points (baseline and weeks 1 through 4), hypothesis tests were performed to test for a differences between baseline and each subsequent time point as well as differences between each time point For data with 3 time points hypothesis tests were performed to test for a differences between baseline and wk 2, wk 2 and wk 4, as well as between baseline and wk 4; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

2. Primary Outcome: Methamphetamine Withdrawal Assessment (MAWA)
Description: The Methamphetamine Withdrawal Assessment (MAWA) is a 13 item questionnaire which measures symptoms of methamphetamine withdrawal on a scale from 0(best score)-4(worst score). The total score ranges from 0(best score)-52(worst score).
Time Frame: Baseline through week 4
Measure: Mean (Standard Deviation); unit: "Units on a scale"
Arm/Group | Methamphetamine Dependent
Number analyzed (Participants) | 6
"Units on a scale" | 20.3 (12.5)
Statistical Analysis 1: Comparison: Methamphetamine Dependent; Means and ranges were computed for continuous baseline(BL)characteristics.For longitudinal data,Proc GLIMMIX in SAS was used to fit a Mixed Model with Random Intercept.For data with 5 time points, hypothesis tests were performed to test for a differences between BL and each subsequent time point as well as differences between each time point. For data with 3 time points, hypothesis tests were performed to test for a differences between BL and wk 2,wk 2and wk 4,as well as between BL and wk 4; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

3. Secondary Outcome: Hamilton Depression Rating Scale (HAM-D) Rating Score
Description: Hamilton Depression rating scale (HAM-D)is a scale that covers 21 symptoms with a total score of 0(best score)-62 (worst score) and a cutoff for moderate depression of 15 or above.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: "Units on a scale"
Arm/Group | Methamphetamine Dependent
Number analyzed (Participants) | 6
"Units on a scale" | 18.5 (13.4)
Statistical Analysis 1: Comparison: Methamphetamine Dependent; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the entire duration of the study 18 months.
Description: No adverse events were identified as this was an observational study.
Arm/Group | Methamphetamine Dependent
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
The small sample size (N=6) is a significant limitation of the current study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes